CLINICAL TRIAL: NCT06528054
Title: TreatmENT of AnastomotiC LeakagE After COLON Cancer Resection: the TENTACLE - Colon Study
Brief Title: TreatmENT of AnastomotiC LeakagE After COLON Cancer Resection
Acronym: TENTACLE-Colon
Status: Not yet recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-3-2500
Record Dates: First submitted 2024-07-24; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Treatment; Anastomotic Leakage; Resection; Colon Cancer
MeSH Terms: conditions — Anastomotic Leak; Colonic Neoplasms | interventions — Mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Development of a model for predicting 90-day mortality and to compare various treatment strategies for anastomotic leakage — The prediction model and comparison of various treatment strategies will be studies when the data is available for analysis.

SUMMARY:
This international multicentre retrospective cohort study aims to research anastomotic leakage after colon cancer resection and has two main objectives:

1. To identify predictive factors associated with 90-day mortality and 90-day Clavien-Dindo grade 4-5 complications amongst patients who developed AL following colon cancer resection and to develop and validate a prediction model for predicting 90-day mortality as well as the co-primary composite endpoint Clavien-Dindo grade 4-5 complications.
2. To explore and compare the effectiveness of various treatment strategies for AL following colon cancer resection, considering patient, tumour, resection and leakage characteristics.

ELIGIBILITY:
Inclusion criteria:

* Aged 18 years or older;
* Surgical resection for primary colon cancer (cT1-4b, N0-2, M0-1) with formation of a primary colonic anastomosis and with or without diverting stoma;
* Postoperative AL defined as: "any clinical, radiological or intraoperative signs of disrupted integrity of the anastomosis. This also includes suspected leaks with any degree of extraluminal air or fluid on CT, perianastomotic abscess, purulent peritonitis without clear anastomotic defect, or any other suspicious condition in which there is no ultimate macroscopic proof of disrupted anastomosis."
* Regarding the type of colon cancer resection, the following patients will also fulfil the inclusion criteria: patients who underwent cytoreductive surgery (CRS) simultaneous with resection of the primary colon cancer with or without hyperthermic intraperitoneal chemotherapy (HIPEC), simultaneous ablations/resections of metastasis, multivisceral resection, emergency resection, patients diagnosed with perforated disease/peritumoral abscess or fistula, and acute obstructions.

Exclusion criteria:

* Surgical resection for benign colon disease;
* Recurrent colon cancer resection;
* Any primary colon malignancy other than adenocarcinoma (e.g. neuroendocrine tumour, gastrointestinal stromal tumour);
* Any clinical condition that does not fulfil the broad definition of AL as used in this study (e.g. only free air on CT that is considered to be compatible with an appropriate postoperative day in the absence of any other clinical signs related to a potential anastomotic leakage)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who developed AL after surgical resection with formation of primary anastomosis for colon cancer (cT1-4bN0-2M0-1).
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
90-day mortality | 90 days after colon cancer resection
  mortality correlated with anastomotic leakage
90-day Clavien-Dindo grade IV - V complications | 90 days after colon cancer resection
  This composite co-primary outcome consists of single-organ failure (i.e. grade IV) and mortality (i.e. grade V)

SECONDARY OUTCOMES:
Time from colon cancer resection to diagnosis of anastomotic leakage | at least one year follow up
Time from colon cancer resection to primary treatment of anastomotic leakage | at least one year follow up
Length of hospital/intensive care unit stay | at least one year follow up
Mortality | 30-day, 90-day and one-year after colon cancer resection
Stoma presence (and if so, type of stoma) | At least one year after colon cancer resection, preferably last date of follow up
Disease status | At least one year after colon cancer resection, preferably at last date of follow up
Number of radiologic and surgical reinterventions | One year after colon cancer resection

CONTACTS AND LOCATIONS:
Overall Officials: Hans de Wilt, Professor, Principal Investigator — Radboud University Medical Center; Pieter Tanis, Professor, Principal Investigator — Erasmus Medical Center

IPD SHARING:
Plan to Share IPD: Undecided
Data may be available upon reasonable request. Only collaborators with appropriate qualifications and pertinent research inquiries are eligible to request access to the data. The principal investigators of the TENTACLE - Colon study will assess the relevance and appropriateness of the request and their verdict is decisive. If data will be transferred, it will solely be conducted under the appropriate ethical and data transfer agreement.

REFERENCES:
- [Derived] Lemmens JMG, Ubels S, Greijdanus NG, Wienholts K, van Gelder MMHJ, Wolthuis A, Lefevre JH, Brown K, Frasson M, Rotholtz N, Denost Q, Perez RO, Konishi T, Rutegard M, Gearhart SL, Pinkney T, Elhadi M, Hompes R, Tanis PJ, de Wilt JHW. TreatmENT of AnastomotiC LeakagE after colon cancer resection: the TENTACLE - Colon study. BMC Surg. 2025 May 15;25(1):213. doi: 10.1186/s12893-025-02954-1. PMID 40375249